CLINICAL TRIAL: NCT02759510
Title: Comparison of Norepinephrine and Phenylephrine in Cesarean Section by Transesophageal Ultrasound
Brief Title: Cardiac Output Changes in Cesarean Section
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Renji-2016035k
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Cardiac Output,Low; Hemodynamic Instability; Obstetrical Complication of Anesthesia
Keywords: cardiac output; norepinephrin; cesarean section
MeSH Terms: conditions — Cardiac Output, Low | interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- phenylephrine (Active Comparator): phenylejphrine (one bolus for 40 ug/ml)
  Interventions: Drug: Phenylephrine
- norepinephrine (Experimental): norepinephrine (one bolus for 2 ug/ml)
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — Hypotension (systolic BP <80% of baseline) will be treated with intravenous boluses of norepinephrine 2 μg.
  Arms: norepinephrine
Drug: Phenylephrine — Hypotension (systolic BP <80% of baseline) will be treated with intravenous boluses of phenylephrine 40 μg.
  Arms: phenylephrine

SUMMARY:
Since 2011, phenylephrine was recommended as the preferred drug to maintain blood pressure in obstetric anesthesia.Phenylephrine, an α adrenoceptor agonist, can induce peripheral vasoconstriction to maintain blood pressure, while reflexly decrease heart rate and result in cardiac output (CO) reduction.Norepinephrine acts not only as an α adrenoceptor receptor agonist, but also as a weaker β adrenergic receptor agonist. It can elevate blood pressure the same asphenylephrine, meanwhile produce positive inotropic effect including increasing heart rate.Thus, the administration of norepinephrine can maintain blood pressue and avoid the decline of CO. The purpose of this study is to evaluate the effect of norepinephrine and phenylephrine on maternal CO in cesarean section by transesophageal echocardiography.

DETAILED DESCRIPTION:
Combined spinal epidural anesthesia (CSEA) is a commonly used anesthetic methods in cesarean section. The main problem of CSEA is hypotension, which will cause maternal nausea and vomiting, reduced uteroplacental blood flow and fetal acidosis. One of the important methods for prevention and treatment of hypotension after CSEA is to give vasoactive drugs.

Since 2011, phenylephrine was recommended as the preferred drug to maintain blood pressure in obstetric anesthesia.Phenylephrine, an α adrenoceptor agonist, can induce peripheral vasoconstriction to maintain blood pressure, while reflexly decrease heart rate and result in cardiac output (CO) reduction.Dyer et al. used bioimpedance technique to analyze the hemodynamic changes in normal pregnant women. A bolus of 80 ug phenylephrine was administrated when maternal mean arterial pressure decreased 20% after CSEA. It was found that cardiac output (CO) decreased significantly (14%) after phenylephrine administrationcompared with the baseline.And the decrease of CO induced by phenylephrine was in a dose dependent.All the studies referred above recruitednormal pregnant women, and the decreased CO did not have an adverse effect on neonatal birth. However, as we all know, the decrease of CO will influence uteroplacental blood, which may lead to adverse results in existed intrauterine distress fetal. All authors of those studies stressed that the decrease of CO induced by phenylephrine may increase the risks of fetal distress or other adverse consequences. So, it is crucial for obstetric anesthesiologist to choose a suitable vasoactive drugs, which can maintain both maternal blood pressure and uteroplacental perfusion in order to keep intrauterine environment steady.

Norepinephrine acts not only as an α adrenoceptor receptor agonist, but also as a weaker β adrenergic receptor agonist. It can elevate blood pressure the same asphenylephrine, meanwhile produce positive inotropic effect including increasing heart rate.Thus, the administration of norepinephrine can maintain blood pressue and avoid the decline of CO. And norepinephrine is superior to phenylephrine in the respect of organ perfusion.

There is little research about the administration of norepinephrine in obstetric anesthesia.Ngan Kee et al.compared phenylephrine (0.57μg/kg/min) with norepinephrine (0.035μg/kg/min) in the treatment of hypotension in obstetric anesthesia. CO monitored by a suprasternal Doppler ultrasound every 5 minutes. CO and heart rate was significantly higher in norepinephrine group than that in phenylephrine group, while peripheral vascular resistance was significantly lower in norepinephrine group than that in phenylephrine group. And the oxygen content in umbilical venous was significantly higher in norepinephrine group, which may be related to the norepinephrine induced lower peripheral vascular resistance and high cardiac output.Monitoring of CO can give a comprehensive understanding of hemodynamics in the pregnant. It enables obstetric anesthesiologist to use liquid expansion rationally and administrate vasoactive agents properly.Although the accuracy of suprasternal Doppler ultrasound was high in that study, the interval of 5min to monitor CO may miss the rapid changes in hemodynamics of pregnant women.In the present study, we will monitor CO continuously by a small diameter (6 mm) transesophageal echocardiography, which can be retained in the patient's esophagus.

The purpose of this study is to evaluate the effect of norepinephrine and phenylephrine on maternal CO in cesarean section by transesophageal echocardiography.Fetal umbilical cord blood, neonatal 1min Apgar score, 5 min Apgar scores and neonatal plasma catecholamine concentrations will be collected to understand the effects of norepinephrine and phenylephrine on fetal.

ELIGIBILITY:
Inclusion Criteria:

1. age >=18 years,<=40 years;
2. height 150-180 cm;
3. weight 55-80 kg;
4. full-term gestation (>36 wk and <41 wk)
5. singleton pregnancy undergoing elective cesarean section under CSEA

Exclusion Criteria:

1. contraindications to spinal anesthesia;
2. patients with any complicated pregnancy;
3. fetal compromise;
4. need of emergency;
5. in labor

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
cardiac output | from baseline (before spinal injection) until 10 minutes after spinal injection

SECONDARY OUTCOMES:
systolic blood pressure | from baseline (before spinal injection) until 10 minutes after spinal injection
heart rate | from baseline (before spinal injection) until 10 minutes after spinal injection
Apgar score | 1 min and 5 min after delivery
Umbilical cord arterial blood pH/BE/Lac | time at delivery
umbilical plasma catecholamine concentration | time at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhou He, MD, Study Chair — Deparment of Anesthesia,South Campus,Renji Hospital,School of Medicine,Shanghai Jiao Tong University,Shanghai,China

IPD SHARING:
Plan to Share IPD: No